CLINICAL TRIAL: NCT00992992
Title: Phase II Study Of Iodine-131 Anti-B1 Antibody Plus CHOP For Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Safety and Efficacy Study of Iodine-131 Anti-B1 Antibody Plus CHOP For Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/005
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP); Tositumomab; Tositumomab and Iodine I-131 tostumomab; Bexxar; Iodine-131 Anti-B1 Antibody; Mantle Cell; radioimmunotherapy
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — tositumomab I-131

ARMS (1):
- Tositumomab and Iodine I 131 Tositumomab followed by CHOP (Experimental): Tositumomab and Iodine I 131 Tositumomab followed by CHOP
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab followed by CHOP

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab followed by CHOP — Patients will receive an infusion of unlabeled Tositumomab (450 mg) followed by an infusion of Tositumomab (35 mg) containing 5 mCi of Iodine-131 (dosimetric dose). Whole body gamma camera scans will be obtained on Day 0; Day 2, 3, or 4; and Day 6 or 7 following the dosimetric dose. Patients will then receive an infusion of unlabeled Tositumomab (450 mg) followed by an infusion of 35 mg Tositumomab containing a patient-specific dose of Iodine-131 calculated to deliver a 75 cGy total body radiation dose (therapeutic dose). Patients who have platelet counts of 100,000-149,000 cells/mm3 will receive 65 cGy; obese patients will be dosed based upon 137% of their lean body mass. Patients will be treated with a thyroid blocking agent 24 hours prior to the dosimetric dose and continuing for 14 days following the therapeutic dose. Approximately 13 weeks following the therapeutic dose, CHOP will be administered every 21 days for a total of 6 cycles.

SUMMARY:
The primary efficacy endpoint of this study is to determine the duration of response of the sequential administration of Iodine-131 Anti-B1 Antibody followed by six cycles of CHOP for patients with previously untreated Mantle Cell Lymphoma (MCL). The secondary efficacy endpoints for this study are to determine the response rate, confirmed response rate, complete response rate, confirmed complete response rate, duration of response for confirmed responders, duration of response for complete responders, duration of response for confirmed complete responders, progression-free survival, time to treatment failure, and the predictive value of detection of minimal residual disease by molecular techniques on response duration. The pharmacokinetic endpoint is to determine the total body residence time of Iodine-131 Anti-B1 Antibody following the dosimetric dose. The safety endpoints are to determine the incidence of adverse experiences, hematologic toxicity, (e.g., nadir, time to nadir, and time to recovery), use of supportive care, percent of patients converting to human anti-murine antibody (HAMA) positivity, the effects of Iodine-131 Anti-B1 Antibody on the growth and function of hematopoietic progenitor cells, and survival of patients with previously untreated MCL treated with Iodine-131 Anti-B1 Antibody followed by six cycles of CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed initial diagnosis of mantle cell non-Hodgkin's lymphoma by histology according to the WHO classification .
* Patients must have Ann Arbor bulky stage II, stage III, or stage IV disease at diagnosis. Bulky stage II disease is defined as a mediastinal mass greater than one-third of the maximum chest diameter, or any other mass greater than or equal to 10 cm in maximum diameter.
* Patients must have less than an average of 25% of the intratrabecular marrow space involved by NHL in bilateral bone marrow biopsy specimens as assessed microscopically at study entry. A unilateral bone marrow biopsy demonstrating <10% involvement with NHL is also adequate.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of paraffin-embedded tissue showing positive reactivity with L26 antibody or immunoperoxidase stains of frozen tissue showing positive reactivity with Anti-B1 Antibody (Coulter Clone) or similar commercially available CD20 antibody or evidence of CD20 positivity by flow cytometry are acceptable evidence of CD20 positivity. This must be performed within 42 days of study entry.
* Patients must have a performance status of at least 60% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
* Patients must have an ANC greater than or equal to 1500 cells/mm3 and a platelet count greater than or equal to 100,000 cells/mm3 within 14 days of study enrollment. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 times the upper limit of normal) and hepatic function (defined as total bilirubin <1.5 times the upper limit of normal and AST <5 times the upper limit of normal) within 14 days of study enrollment.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be greater than or equal to 2.0 x 2.0 cm by computerized tomography scan.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.
* Patients must have a cardiac left ventricular ejection fraction of greater than or equal to 50% by ventriculography or echocardiogram.

Exclusion Criteria:

* Patients who have received prior chemotherapy, biologic therapy, steroids, or radiation therapy as treatment for their MCL
* Patients with active obstructive hydronephrosis
* Patients with serious illness that would preclude evaluation
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for 5 years
* Patients with known HIV infection
* Patients who are HAMA positive
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or breastfeeding. Males and females must agree to use a contraceptive method while on study and for 6 months after receiving Iodine-131 Anti-B1 Antibody.
* Patients with active infection requiring IV anti-infectives at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-06-28 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20064

REFERENCES:
- [Background] Zelenetz AD, Popplewell LL, Noy A, Horner TJ, Lin TS, Donnelly G, Sgouros G, Rijo I, Divgi CR. Phase 2 Study of Iodine-131 Tositumomab Plus Chemotherapy in Patients With Previously Untreated Mantle-Cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2020 Nov;20(11):749-756.e1. doi: 10.1016/j.clml.2019.04.010. Epub 2019 Apr 29. PMID 32800518

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodine I-131 Tositumomab + CHOP: Participants (par.) with previously untreated mantle cell lymphoma (MCL) were dosed with iodine I-131 tositumomab in two phases, followed by six cycles (21 days per cycle) of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP). In the first phase (dosimetric dose), par. received an infusion of unlabeled tositumomab (450 milligrams [mg]) over the course of 60 minutes, followed by a 30-minute infusion of tositumomab (35 mg) containing 5 millicurie (mCi) of iodine-131. In the second phase (therapeutic dose), par. received a 60-minute infusion of tositumomab (450 mg), followed by a 30-minute infusion of 35 mg tositumomab containing a participant-specific dose of iodine-131. This dose was calculated based on the dosimetric dose results to deliver a total body radiation dose of 75 centigray (cGy).
Period: Overall Study
Arm/Group | Iodine I-131 Tositumomab + CHOP
Started | 25
Completed | 0
Not Completed | 25
Not completed — Lost to Follow-up | 3
Not completed — Death | 16
Not completed — GlaxoSmithKline Closed the Study | 2
Not completed — Sponsor Closed the Study | 4

BASELINE CHARACTERISTICS:
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 23
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Unconfirmed Response (Complete Response, Complete Response Unconfirmed, and Partial Response)
Description: Participants with response include those with complete response (CR: complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms), complete response unconfirmed (CRu: CR, with one of the following: residual lymph node mass >1.5 centimeters [cm] that has regressed by more than 75% in the sum of the product of the diameters or indeterminate bone marrow), or partial response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population: all participants who received any iodine I-131 tositumomab or CHOP treatment. Only those participants evaluable for response (those with at least one response assessment) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
Participants
  CR | 14
  CRu | 2
  PR | 5
Statistical Analysis 1: Comparison: Iodine I-131 Tositumomab + CHOP; Test type: Superiority or Other; Percentage of participants = 56, 95% CI 2-sided [37 to 75] — The estimated value reflects the percentage of participants with unconfirmed complete response (CR)
Statistical Analysis 2: Comparison: Iodine I-131 Tositumomab + CHOP; Test type: Superiority or Other; Percentage of participants = 8, 95% CI 2-sided [0 to 19] — The estimated value reflects the percentage of participants with unconfirmed complete response unconfirmed (CRu)
Statistical Analysis 3: Comparison: Iodine I-131 Tositumomab + CHOP; Test type: Superiority or Other; Percentage of participants = 20, 95% CI 2-sided [4 to 36] — The estimated value reflects the percentage of participants with unconfirmed partial response

2. Secondary Outcome: Number of Participants With the Indicated Confirmed Response (Confirmed Complete Response, Complete Response Unconfirmed, and Partial Response)
Description: A confirmed response is defined as a response that was confirmed by two separate response evaluations occurring at least 4 weeks apart. Participants with a confirmed response include those with complete response (CR: complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms), complete response unconfirmed (CRu: CR, with one of the following: residual lymph node mass >1.5 cm that has regressed by more than 75% in the sum of the product of the diameters or indeterminate bone marrow), or partial response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions). The individual rows for confirmed CR, confirmed CRu, and confirmed PR represent confirmation of the same response. For example, a confirmed CR indicates that a CR was followed by another CR at least 4 weeks later.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only those participants evaluable for response (those with at least one response assessment) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 22
Participants
  Confirmed CR | 11
  Confirmed CRu | 2
  Confirmed PR | 3

3. Secondary Outcome: Duration of Response for All Confirmed Responders (CR + CRu + PR)
Description: Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms. Complete response unconfirmed (CRu) is defined as CR, with one of the following: residual lymph node mass >1.5 cm that has regressed by more than 75% in the sum of the product of the diameters or indeterminate bone marrow. Partial response (PR) is defined as a >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions. For participants with CR, CRu, or PR, duration of response is defined as the time from the first documented response to the first documented progression.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only those participants (par.) with a confirmed CR, CRu, or PR were analyzed. The number of par. analyzed represents the par. with a confimed CR, CRu, or PR who also had the same response or a better response as confirmation (for example, a par. with an initial CRu and a subsequent CR has been included in the analysis).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 19
Months | 29.8 [15.8 to NA] — There were too few events of response to calculate an upper limit of the confidence interval.

4. Secondary Outcome: Duration of Response for All Unconfirmed Responders (CR + CRu + PR)
Description: Complete response (CR) is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms. Complete response unconfirmed is defined as CR, with one of the following: residual lymph node mass >1.5 cm that has regressed by more than 75% in the sum of the product of the diameters or indeterminate bone marrow. Partial response (PR) is defind as a >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions. Duration of response is defined as the time from the first documented response to the first documented progression.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only those participants with an unconfirmed response (CR, CRu, or PR) were analyzed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 21
Months | 29.8 [15.8 to NA] — There were too few events of response to calculate an upper limit of the confidence interval.

5. Secondary Outcome: Duration of Response for Unconfirmed Complete Responders
Description: Complete response is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms. Duration of response is defined as the time from the first documented response to the first documented progression.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only those participants with unconfirmed CR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 14
Months | 31.8 [15.8 to NA] — There were too few events of response to calculate an upper limit of the confidence interval.

6. Secondary Outcome: Duration of Response for Confirmed Complete Responders
Description: Complete response is the complete disappearance of all detectable clinical and radiographic evidence of disease and the disappearance of all disease-related symptoms. A confirmed response is defined as a response that was confirmed by two separate response evaluations occurring at least 4 weeks apart. Duration of response is defined as the time from the first documented response to the first documented progression.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only those participants with confirmed CR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 11
Months | 54.0 [15.5 to NA] — There were too few events of response to calculate an upper limit of the confidence interval.

7. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the start of treatment (i.e., the dosimetric dose) to the first documented disease progression or death. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must have been greater than 2 centimeters (cm) in diameter by radiographic evaluation or greater than 1 cm in diameter by physical examination.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Months | 27.6 [17.1 to 39.1]

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from the date of the dosimetric dose to the first occurrence of treatment withdrawal, decision to seek additional therapy, study removal, disease progression, alternative therapy, or death.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Months | 20.2 [15.2 to 34.2]

9. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAEs are defined as those events that were fatal or immediately life-threatening, and those events that resulted in hospitalization; prolonged an existing hospitalization; resulted in disability; or was a congenital anomaly. Refer to the general AE/SAE module for a complete list of all AEs and SAEs.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Participants
  Any AE | 25
  Any SAE | 19

10. Secondary Outcome: Mean Nadir Value for Absolute Neutrophil Count (ANC)
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. ANC is a measure of the number of neutrophil granulocytes present in the blood. Neutrophils are a type of white blood cell that fights infection.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only 24 participants had ANC data available.
Measure: Mean (Standard Deviation); unit: 1000 cells/millimeters cubed (mm^3)
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
1000 cells/millimeters cubed (mm^3) | 1.8 (0.93)

11. Secondary Outcome: Mean Nadir Value for Hemoglobin
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Hemoglobin is the iron-containing oxygen-transport metalloprotein in the red blood cells.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only 24 participants had hemoglobin data available.
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
grams/deciliter (g/dL) | 11.2 (1.51)

12. Secondary Outcome: Mean Nadir Values for Platelets and White Blood Cell (WBC) Count
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Platelets and WBCs are types of blood cells.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only 24 participants had platelet and WBC data available.
Measure: Mean (Standard Deviation); unit: 1000 cells/microliter
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
1000 cells/microliter
  Platelet count | 80.7 (54.18)
  WBC count | 2.8 (1.30)

13. Secondary Outcome: Time to Nadir for the Indicated Hematology Parameters
Description: Hematology parameters include ANC (calculated), hemoglobin, platelet count, and WBC count. Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Time to nadir is defined as the time from Baseline to the time the lowest value recorded following the therapeutic dose.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only 24 participants had data available.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
Days
  ANC | 42.9 (5.93)
  Hemoglobin | 62.1 (41.35)
  Platelet count | 45.7 (31.51)
  WBC count | 55.9 (29.43)

14. Secondary Outcome: Time to Recovery From the Indicated Hematology Parameters
Description: Hematology parameters include ANC (calculated), hemoglobin, platelet count, and WBC count. Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Time to recovery to Baseline for the indicated hematologic parameters is defined as the time required for recovery from nadir values to Baseline values.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population. Only 24 participants had data available.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 24
Days
  ANC | 49.5 [44.0 to 55.0]
  Hemoglobin | 84.0 [41.0 to 115.0]
  Platelet count | 43.5 [42.0 to 50.0]
  WBC count | 53.0 [50.0 to 84.0]

15. Secondary Outcome: Number of Participants Negative for Human Anti-Murine (Mouse) Antibody (HAMA) at Screening Who Converted to HAMA Positivity or Remained Negative During the Course of the Study
Description: The number of participants who developed human anti-murine (mouse) anibodies (HAMA) after treatment was measured. Conversion to HAMA positivity is relative to Screening (participants were evaluable for HAMA analysis if they were HAMA negative at Screening).
Time Frame: Screening; at Week 7, Week 13, then every 6 months until disease progression or death (up to 143 months)
Population: ITT-Exposed Population. Only those participants evaluable for HAMA were analyzed.
Measure: Number; unit: Participants
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 23
Participants
  Positive | 10
  Negative | 13

16. Secondary Outcome: Number of Participants With an Adverse Event of Cytopenia
Description: The effects of iodine I-131 tositumomab on the growth and function of hematopoietic progenitor cells was measured as the number of participants who had cytopenia. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Participants
  Thrombocytopenia | 3
  Pancytopenia | 1

17. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment to the date of death from any cause.
Time Frame: Every 13 weeks up to 2 years, or every 6 months until disease progression or death (average of 77.8 months)
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Iodine I-131 Tositumomab + CHOP
Number analyzed (Participants) | 25
Months | 83.1 [56.5 to 121.6]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until 4 weeks following the last cycle of CHOP, or until administration of alternative therapy, whichever came first (average of 77.8 months).
Arm/Group | Iodine I-131 Tositumomab + CHOP
Serious Adverse Events (participants affected / at risk) | 19/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iodine I-131 Tositumomab + CHOP (N=25)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iodine I-131 Tositumomab + CHOP (N=25)
Fatigue (General disorders) | 21
Pyrexia (General disorders) | 9
Chills (General disorders) | 4
Pain (General disorders) | 4
Chest discomfort (General disorders) | 3
Mucosal inflammation (General disorders) | 3
Asthenia (General disorders) | 2
Early satiety (General disorders) | 2
Local swelling (General disorders) | 2
Oedema peripheral (General disorders) | 2
Chest pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema (General disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Inguinal hernia (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 10
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 3
Burning sensation (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Platelets <50000 cells/millimeters cubed (mm^3) (Investigations) | 10
WBC < 2000 cells/mm^3 (Investigations) | 10
Absolute neutrophil count (CALC) < 1000 cells/mm^3 (Investigations) | 6
Hemoglobin < 8.0 grams per deciliter (g/dL) (Investigations) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6
Folliculitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Goitre (Endocrine disorders) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 2
Antibody test abnormal (Investigations) | 1
Blood glucose increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Hypotension (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Halo vision (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cardiac septal defect (Congenital, familial and genetic disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.